CLINICAL TRIAL: NCT04005651
Title: Post-Market Follow-up Clinical Trial to Investigate Safety and Efficacy of a Trifocal Intraocular Lens (IOL) POD L GF In Comparison With a Multifocal (TECNIS Symfony® Extended Range of Vision IOL) and a Monofocal (AcrySof® IQ Monofocal IOL)
Brief Title: Safety and Efficacy of a Trifocal Intraocular Lens (IOL) POD L GF in Comparison With a Multifocal and a Monofocal IOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beaver-Visitec International, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHY1804
Record Dates: First submitted 2019-06-26; First posted 2019-07-02 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Aphakia, Postcataract; Cataract; Eye Disease
MeSH Terms: conditions — Aphakia, Postcataract; Cataract

STUDY DESIGN:
Intervention Model Description: Approximately 150 subjects will be implanted bilaterally with 50 subjects implanted with the POD L GF lenses, 50 subjects implanted with the Symfony® intraocular lenses, and 50 subjects implanted with the AcrySof® monofocal lenses. The objective is to complete approximately 141 subjects through 12 month post-operative follow-up (~47 subjects in each cohort).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- POD L GF (Experimental): Approximately 50 subjects who are scheduled for multifocal IOL implantation and enrolled in the study will be randomized into the POD L GF arm. Subjects will be implanted bilaterally with the European Conformity (CE) marked POD L GF trifocal IOL and assessed according to the study visit schedule.
  Interventions: Device: POD L GF IOL
- Symfony® (Active Comparator): Approximately 50 subjects who are scheduled for multifocal IOL implantation and enrolled in the study will be randomized into the Symfony arm. Subjects will be implanted bilaterally with the CE marked TECNIS Symfony® IOL and assessed according to the study visit schedule.
  Interventions: Device: Symfony® IOL
- AcrySof® (Active Comparator): Approximately 50 subjects who are scheduled for monofocal IOL implantation and enrolled in the study will be placed in the AcrySof® arm. Subjects will be implanted bilaterally with the CE marked AcrySof® IQ monofocal IOL and assessed according to the study visit schedule.
  Interventions: Device: AcrySof® IOL

INTERVENTIONS:
Device: POD L GF IOL — Cataractous lens will be removed in the study eyes and the POD L GF IOL will be implanted in the capsular bag
  Arms: POD L GF
Device: Symfony® IOL — Cataractous lens will be removed in the study eyes and the Symfony® IOL will be implanted in the capsular bag
  Arms: Symfony®
Device: AcrySof® IOL — Cataractous lens will be removed in the study eyes and the AcrySof® IOL will be implanted in the capsular bag
  Arms: AcrySof®

SUMMARY:
The objectives of the Post-Market Follow-up (PMCF) clinical investigation are to determine the safety and performance of a hydrophobic trifocal intraocular lens POD L GF in comparison with two comparator lenses: another multifocal intraocular lens (Johnson & Johnson TECNIS Symfony® Extended Range of Vision IOL); and a monofocal intraocular lens (Alcon AcrySof® IQ Monofocal IOL) through one year of post-operative assessments.

DETAILED DESCRIPTION:
This is a prospective, multicenter, randomized, active controlled comparative binocular Post Market Follow-up (PMCF) clinical study to demonstrate safety and efficacy between the trifocal intraocular lens POD L GF and the Johnson & Johnson TECNIS Symfony® Extended Range of Vision IOL and the Alcon AcrySof® IQ Monofocal IOL.

Patients who are scheduled to undergo cataract extraction in one or both eyes and posterior chamber intraocular lens implants may be screened for eligibility in the study and, if eligible, complete a pre-operative screening visit. Both eyes of subjects who are eligible to receive the POD L GF IOL or the Johnson & Johnson TECNIS Symfony® Extended Range of Vision IOL must be eligible to receive bilateral multifocal IOL implants. Both eyes of subjects who are eligible to receive the Alcon AcrySof® IQ Monofocal IOL must be eligible to receive bilateral monofocal IOL implants.

At the time of the first eye surgery, the subjects to be implanted with either the POD L GF (test) IOL or the Johnson & Johnson TECNIS Symfony® Extended Range of Vision (comparator) IOL will be randomized to receive either the test or comparator IOL in a 1:1 ratio. In addition, 50 subjects will be implanted with the Alcon AcrySof® IQ Monofocal IOL. All subjects will undergo bilateral IOL implantation and will receive the same brand of lenses in each eye. Second eye implantations will be delayed until 1 to 30 days after the first eye implantation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults ages 45 or older on the day of screening who have cataract(s) in one or both eyes
* Capability to understand and sign an Ethics Committee (EC) approved informed consent form and privacy authorization
* Corrected visual acuity projected by potential acuity meter (PAM) testing or other potential visual acuity test procedure to be better than 20/32 after intraocular lens implantation
* Clear intraocular media other than cataract
* Calculated IOL power is within the range of the study IOLs
* Dilated pupil size large enough to visualize IOL axis markings postoperatively
* Willing and able to conform to the study requirements

Exclusion Criteria:

* Subjects with diagnosed degenerative visual disoerders (e.g., macular degeneration or other retinal or optic disorders) that are predicted to cause future acuity losses to a level of 20/30 or worse
* Subjects with age-related macular degeneration (AMD) suspicious eyes as determined by optical coherence tomography (OCT) examination
* Subjects who may be expected to require retinal laser treatment during the course of the study or at a greater risk of developing cystoid macular edema
* Greater than 1 diopter of pre-operative corneal astigmatism or any irregular astigmatism
* Previous intraocular or corneal surgery
* Traumatic cataract
* History or presence of macular edema
* Pregnant,lactating or, if able to bear children, unwilling to use medically acceptable birth control over the course of the study
* Concurrent or previous (within 30 days) participation in another drug or device investigation
* Instability of keratometry or biometry measurements
* Ocular hypertension or glaucoma
* Significant dry eye
* Unsuitable for study participation for any other reason, as determined by Investigator's clinical judgement (reason to be documented on eCRF)

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-05-30 (Actual); Primary Completion 2022-07-27 (Actual); Study Completion 2022-11-29 (Actual)

PRIMARY OUTCOMES:
CDVA in first implanted eyes | Day 120-180 both eyes
  Photopic monocular logMAR corrected distance visual acuity (CDVA) in first implanted eyes at Visit 4
DCIVA in first implanted eyes | Day 120-180 both eyes
  Photopic monocular logMAR intermediate visual acuity with distance correction (DCIVA) in first implanted eyes at Visit 4
DCNVA in first implanted eyes | Day 120-180 both eyes
  Photopic monocular logMAR near visual acuity with distance correction (DCNVA) in first implanted eyes at Visit 4

SECONDARY OUTCOMES:
UDVA at Visits 3A, 3B, 4, and 5 | Day 30-60 post first eye (3A), day 30-60 post second eye (3B), day 120-180 both eyes (4), day 330-420 both eyes (5)
  Photopic monocular logMAR uncorrected distance visual acuity (UDVA)
UIVA at Visits 3A, 3B, 4, and 5 | Day 30-60 post first eye (3A), day 30-60 post second eye (3B), day 120-180 both eyes (4), day 330-420 both eyes (5)
  Photopic monocular logMAR uncorrected intermediate visual acuity (UIVA)
UNVA at Visits 3A, 3B, 4, and 5 | Day 30-60 post first eye (3A), day 30-60 post second eye (3B), day 120-180 both eyes (4), day 330-420 both eyes (5)
  Photopic monocular logMAR uncorrected near visual acuity (UNVA)
CDVA at Visits 3A, 3B, 4, and 5 | Day 30-60 post first eye (3A), day 30-60 post second eye (3B), day 120-180 both eyes (4), day 330-420 both eyes (5)
  Photopic monocular logMAR corrected distance visual acuity (CDVA)
DCIVA at Visits 3A, 3B, 4, and 5 | Day 30-60 post first eye (3A), day 30-60 post second eye (3B), day 120-180 both eyes (4), day 330-420 both eyes (5)
  Photopic monocular logMAR intermediate visual acuity with distance correction (DCIVA)
DCNVA at Visits 3A, 3B, 4, and 5 | Day 30-60 post first eye (3A), day 30-60 post second eye (3B), day 120-180 both eyes (4), day 330-420 both eyes (5)
  Photopic monocular logMAR corrected near visual acuity with distance correction (DCNVA)
Quality of Vision Questionnaire (QoV) quality of vision at Visit 4 | Day 120-180 both eyes
  Quality of vision based on response to each question in the Quality of Vision (QoV) questionnaire at Visit 4. Answer is a choice of 4 options, the first being the least and the fourth being the most based on question type, i.e. "never" to "very often" or "not at all" to "severe".
Near Activity Visual Questionnaire (NAVQ) quality of vision at Visit 4 | Day 120-180 both eyes
  Quality of vision based on response (choice of 0-3 with 0 meaning no difficulty and 3 meaning extreme difficulty) to each question in the Near Activity Visual Questionnaire (NAVQ) at Visit 4.

OTHER OUTCOMES:
Safety Endpoint: Rates of AEs (Adverse Events) | Enrollment (Day -30 to -1) through study exit or Visit 5 (Day 330 to 420 both eyes), whichever comes first
  Rates of posterior chamber IOL adverse events compared to the ISO Safety and Performance Endpoint (SPE) rates as described in International Organization for Standardization (ISO) 11979-7
Safety Endpoint: Optical and Visual Symptoms Assessed with NAVQ | Visit 4 (Day 120 to 180 both eyes)
  Subject questionnaire frequency of optical and visual symptoms as reported in NAVQ
Safety Endpoint: Optical and Visual Symptoms Assessed with QoV questionnaire | Visit 4 (Day 120 to 180 both eyes)
  Subject questionnaire frequency of optical and visual symptoms as reported in QOV questionnaire
Safety Endpoint: Secondary Surgical Interventions | Operative Visit (Day 0) through study exit or Visit 5 (Day 330 to 420 both eyes), whichever comes first
  Rates of device-related secondary surgical interventions related to the POD L GF trifocal IOL
Safety Endpoint: Serious Adverse Events | Day 330 to 420 both eyes
  The rate of serious adverse events related to teh POD L GF trifocal IOL in first implanted eyes through Visit 5

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Pagnoulle, Study Director — PhysIOL s.a.
Locations (5):
- OphtALLIANCE Clinique Jules Verne, Nantes, France
- Germany (3):
  - Augenklinik Ahaus, Ahaus
  - Internationale Innovative Ophthalmochirgie, Düsseldorf
  - Augentagesklinik Rheine, Rheine
- IOA Madrid Innova Ocular, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No